CLINICAL TRIAL: NCT04329091
Title: Implications of Anesthetics on Sleep Consolidation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of participant recruitment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB19-1442
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Sleep
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexmedetomidine Arm (Experimental): Dexmedetomidine: Administration of a 0.5 mcg/kg bolus followed by an infusion of 0.5-0.7 mcg/kg/hr, titrated up by 0.1 mcg every 1 minute until the subject spontaneously closes his or her eyes. When the subject spontaneously closes his or her eyes the infusion continues for 90 minutes from that point.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — All subjects will receive Dexmedetomidine to induce sedation between their pre-sedation and post-sedation perceptual learning tests.
  Other Names: Precedex

SUMMARY:
Sleep leads to consolidation of learning in humans, restoring memories that were forgotten over a waking day and protecting memories against future forgetting. Although theories of consolidation have linked sleep spindles seen on electroencephalography to consolidation due to their putative role in hippocampal transfer to the neocortex (Antony et al, 2019; Antony & Paller, 2017), spindles have not yet been linked to consolidation of perceptual learning or generalized learning. Prior research by a collaborator on this project has shown that sleep specifically aids in the consolidation of generalized perceptual learning of speech (Fenn, Nusbaum, & Margoliash, 2003). Subjects show a 10-point reduction in performance after a waking retention period, while no loss is found after a retention period containing sleep (Fenn et al., 2003).

Various measurable activities in the brain are associated with memory consolidation during sleep. This project intends study the effect of dexmedetomidine on memory consolidation during sleep

Hypothesis 1 The gain in perceptual learning after a 90 minute natural sleep nap will also occur after 90 minutes of a sufficient dose of IV dexmedetomidine to replicate sleep. This result would suggest that consolidation can occur under this anesthetic state of consciousness.

Hypothesis 2 The number and quality of sleep spindles seen on EEG in subjects administered dexmedetomidine will correlate with this gain in perceptual learning. This result would suggest that biomimetic sleep spindles are sufficient for producing memory consolidation.

Only those subjects capable of giving their own consent will be considered for this study.

The study will enroll 20 healthy subjects for this study between the ages of 18 and 35.

All volunteers will be fit and healthy, meeting the American Society of Anesthesiologists (ASA) physical status classification ASA 1 (normal healthy subjects) and ASA 2 (stable chronic condition) and of normal body habitus. Prior to the study enrollment, each volunteer will sign an informed consent form. A standard anesthetic medical history will be taken in addition to performing a focused standard pre-anesthetic physical examination in order to rule out active and chronic medical problems.

ELIGIBILITY:
Primary Inclusion Criteria for "Healthy" volunteers

* Age between 18-35
* Native English speaking
* No hearing or speech difficulties
* No psychiatric, neurologic, or sleep disorders
* No chronic medical conditions, as reflected below under Primary Exclusion Criteria and above in 'Medical History'
* Non-smokers (within 3 months)
* Non-users of recreational or illicit drugs (including marijuana)
* Must be willing and able to pass the drug tests (no psychoactive substances), no ingestion of alcohol or sleep-altering drugs for the 48 hours prior to the study session.
* Normal weight

Primary Exclusion Criteria for "Healthy" volunteers

* Speech difficulties/disorders
* Hearing difficulties (including occluded or infected ear canals)
* Current hairstyles that do not allow the high-density EEG cap to make contact with the scalp (e.g., individuals with hair extensions, braids, dreadlocks or hairstyles that restrict the ability of electrodes to touch the scalp)
* Metal on/in/near their heads (including jewelry) that cannot be removed for the duration of the study
* Metal implants
* Serious abusers of alcohol or caffeine.
* Existing or suspected psychological or neurological disorders
* Pregnancy or suspected pregnancy (urine pregnancy test at visit 2)
* Chronic or transient (e.g., jet lag) problems with sleep; suspected sleep disorder
* Abnormal sleep habits, such as:

  * Sleeping less than 5 hours each night
  * Going to sleep before 8:00 PM or after 2:00 AM on a regular basis
  * Waking up before 5:00 AM or after 10:00 AM on a regular basis.
* Currently taking medications that regulate blood pressure; a history of high blood pressure, diabetes or stroke
* Chronic smokers
* Current use of aspirin, or other medications which increase bleeding, prior to the study session.
* Known drug allergies to anesthetics or a history of an adverse reaction to anesthesia.
* Known allergy to adhesives or electrode gel
* Medication that alters sleep, cognitive function, or both

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Clebone, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine Arm
Started | 9 (First subject enrolled)
Completed | 4 (Last subject follow up.)
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Dexmedetomidine Arm
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 9
Memory consolidation [Count of Participants; unit: Participants] — Population: No data was collected or analyzed

OUTCOME MEASURES:

1. Primary Outcome: Perceptual Learning Protocol
Description: Subjects are tested in the morning for word recognition on hard-to-understand speech, then trained on this speech (never hearing the same words twice) which produces about 20 percentage points of improvement. After sedation subjects are re-tested. During the morning, afternoon and evening post-tests, subjects will be tested on new spoken words. At each time point where the perceptual learning protocol is administered the number of words correctly perceived out of 50 will be measured.
Time Frame: 1 day
Population: Study terminated, no data was collected.
Arm/Group | Dexmedetomidine Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Dexmedetomidine Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04329091/Prot_SAP_001.pdf